CLINICAL TRIAL: NCT03459651
Title: Investigation of the Role of Turner Syndrome on Approximate Number Sense
Brief Title: Effect of Turner Syndrome on Number Sense
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator elected to end the study.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Joseph Michael Baker, Instructor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 092883
Record Dates: First submitted 2018-02-27; First posted 2018-03-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Turner Syndrome
Keywords: numeracy; number sense
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANS training (Experimental)
  Interventions: Behavioral: ANS training

INTERVENTIONS:
Behavioral: ANS training — In-home computer-based ANS training

SUMMARY:
This study evaluates approximate number sense (ANS) in children, adolescents, and adult women with Turner syndrome compared to age-matched healthy peers. One primary aim of this project is to assess the effectiveness of an online ANS training tool in enhancing complex mathematics ability. Participants will undergo weekly training sessions in their own home. Half of the participants will complete 2 training sessions a week for 8 weeks, and the second half will complete 1 training session for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents, and adult women with Turner syndrome.
* Healthy controls.
* Normal or corrected to normal vision.

Exclusion Criteria:

* Major psychiatric or developmental disorder (e.g., bipolar disorder, major depression, psychotic disorders, intellectual disability, autism spectrum disorder).
* Chemical dependency
* Currently taking the following medications: antidepressant, antipsychotic, and anti-seizures drugs.

Ages: 6 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
Single and multiple-operand addition and subtraction accuracy | 8 weeks
  Task accuracy calculated as the percentage of trials answered correctly.
Single and multiple-operand addition and subtraction response time | 8 weeks
  Average amount of time, in seconds, required to answer each question on the task.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Interdisciplinary Brain Sciences Research, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for the primary outcome measures may be made available upon reasonable request.